CLINICAL TRIAL: NCT01499433
Title: Prospective, Open-label Study of the Efficacy and Safety of Caspofungin for the Treatment of Invasive Pulmonary Aspergillosis Underlying Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of Caspofungin for Invasive Pulmonary Aspergillosis Underlying Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Feng Ye, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IISP# 39758
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Invasive Pulmonary Aspergillosis; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Pulmonary Disease, Chronic Obstructive | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- caspofungin (Experimental)
  Interventions: Drug: caspofungin

INTERVENTIONS:
Drug: caspofungin — Caspofungin injection, intravenously administered, loading dose at 70mg qd for the first 24hrs, maintenance dose at 50mg qd for the following 20 days
  Other Names: brand name:Cancidas

SUMMARY:
The investigators propose to study the efficacy and safety of three-week antifungal therapy with caspofungin in hospitalized patients with proven or probable IPA underlying chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Recently, there has been increasing appreciation of chronic obstructive pulmonary disease (COPD) as an important risk factor of invasive pulmoanry aspergillosis (IPA). However, clinical data on the morbidity and mortality of IPA underlying COPD as well as the efficacy and safety of antifungal treatment in such subset of patient population is very limited. In clinical pratice, capofungin is often used as primary antifungal therapy for IPA, especially in patients with impaired renal function. Based on this data, the investigators propose to study the efficacy and safety of three-week antifungal therapy with caspofungin in hospitalized patients with proven or probable IPA underlying COPD.

ELIGIBILITY:
Inclusion Criteria:

* Proven invasive pulmonary aspergillosis
* Probable invasive pulmonary aspergillosis
* Hospitalized in respiratory wards
* Not having received an empirical antifungal therapy for 72h before inclusion

Exclusion Criteria:

* A history of allergy to echinocandins
* Severe renal failure, severe hepatic insufficiency
* Inadequately treated bacterial infection
* Documented HIV infection
* Status of pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Global response (defined as both clinical and microbiologic success) at the end of intravenous therapy | At end of intravenous treatment(three week)
  The primary objective is to investigate the clinical efficacy of 3-week treatment with caspofungin as either primary or salvage antifungal therapy for IPA underlying COPD.

SECONDARY OUTCOMES:
Assessment of Safety of Caspofungin for IPA Underlying COPD | at the time of enrollment, weekly during therapy, and 1 week after the end of therapy.
  Safety evaluation : Laboratory examinations are performed; Number of participants with adverse events are recorded.
Global response to 2-week caspofungin therapy | 2 week
Factors such as severity of COPD, exposure to systemic corticosteroids,extended-spectrum antibiotics et al. affecting patients' response to caspofungin therapy | 3 week
  Assessment of factors such as severity of COPD, exposure to systemic corticosteroids,extended-spectrum antibiotics,malnutrition or diabetes affecting patients' response to caspofungin therapy
Clinical response at Day 7 of treatment | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ye, MD, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Diseases, Guangzhou, Guangdong, China